CLINICAL TRIAL: NCT04905108
Title: Randomized Study of Safety and Effectiveness of Corneal Collagen Crosslinking Using Two Different Riboflavin Administration Protocols
Brief Title: Transepithelial (Epi-on) Corneal Collagen Crosslinking to Treat Keratoconus and Corneal Ectasia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cornea and Laser Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TE-CXL-002
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Keratoconus; Corneal Ectasia
Keywords: keratoconus; corneal ectasia; collagen crosslinking; riboflavin; crosslinking; corneal crosslinking
MeSH Terms: conditions — Keratoconus | interventions — Riboflavin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Riboflavin drop every 2 minutes (Active Comparator): Administration of one drop of Riboflavin every 2 minutes during UV exposure
  Interventions: Drug: Riboflavin
- Riboflavin drop every 10 minutes (Active Comparator): Administration of one drop of Riboflavin every 10 minutes during UV exposure
  Interventions: Drug: Riboflavin

INTERVENTIONS:
Drug: Riboflavin — Administration of riboflavin one drop every 2 minutes during UVA exposure
  Arms: Riboflavin drop every 10 minutes
Drug: Riboflavin — Administration of riboflavin one drop every 10 minutes during UVA exposure
  Arms: Riboflavin drop every 2 minutes

SUMMARY:
Corneal collagen crosslinking (CXL) has been demonstrated as an effective method of reducing progression of both keratoconus and corneal ectasia after surgery, as well as possibly decreasing the steepness of the cornea in these pathologies. Transepithelial crosslinking in which the epithelium is not removed has been proposed to offer a number of advantages over traditional crosslinking including an increased safety profile by reducing the risk for infection and scarring, faster visual recovery and improved patient comfort in the early postoperative healing period.

DETAILED DESCRIPTION:
The objective of this randomized study is to investigate the difference between two regimens of transepithelial crosslinking. The study will compare two riboflavin dosing regimens during the crosslinking procedure. The primary objective of this study is to evaluate the safety and efficacy of transepithelial corneal collagen crosslinking performed with two different riboflavin administration protocols during the UVA portion of the procedure. Safety and efficacy outcomes will then be compared between the treatment groups. In particular, the two groups will be compared with regard to their efficacy in reducing corneal curvature. Secondary outcomes will include visual acuity. Safety assessments will include a tabulation of adverse events, patient symptoms, loss of visual acuity, changes in endothelial cell density, and slit lamp examination.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age or older
* Having a diagnosis of keratoconus or corneal ectasia after corneal refractive surgery (e.g., LASIK, photorefractive keratectomy [PRK])
* Presence of central or inferior steepening on the Pentacam map
* Axial topography consistent with keratoconus or post-surgical corneal ectasia
* Contact lens wearers only: Removal of contact lenses for the required period of 1 week prior to the screening refraction
* Signed written informed consent
* Willingness and ability to comply with schedule for follow-up visits

Exclusion Criteria:

* Eyes classified as either normal, atypical normal, or keratoconus suspect on the severity grading scheme
* Corneal pachymetry measuring 300 microns or less at the thinnest point measured by Pentacam in the eye(s) to be treated
* Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye for future complications, for example:

  1. History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, corneal melt, corneal dystrophy, etc.)
  2. Clinically significant corneal scaring in the CXL treatment zone
* A history of chemical injury or delayed epithelial healing in the eye(s) to be treated
* Pregnancy (including plan to become pregnant) or lactation during the course of the study
* A known sensitivity to study medications
* Patients with nystagmus or any other condition that would prevent a steady gaze during the CXL treatment or other diagnostic tests
* Patients with a current condition that,in the investigator's opinion, would interfere with or prolong epithelial healing

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Maximum keratometry | 12 months
  The change in maximum keratometry (Kmax) from baseline will be evaluated at 12 months for all eyes randomized in group 1 and group 2.

SECONDARY OUTCOMES:
Mean keratometry | 1 year
  The change in mean keratometry (Mean K) from baseline will be evaluated at 12 months for all eyes randomized in group 1 and group 2.

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Hersh, MD, Study Director — Cornea and Laser Eye Institute - Hersh Vision Group; Steven A Greenstein, MD, Principal Investigator — Cornea and Laser Eye Institute - Hersh Vision Group
Locations (1):
- Cornea and Laser Eye Institute, Hersh Vision Group, Teaneck, New Jersey, United States